CLINICAL TRIAL: NCT06190509
Title: Candi5V01 A FTIH Phase I/II Randomized and Controlled Study to Test Safety, Immunogenicity and Preliminary Efficacy of a Pentavalent Bioconjugate Vaccine (Candi5V) Against Candida in Women With Recurrent Vulvovaginal Candidiasis.
Brief Title: Assessing the Safety, Immune Response, and Early Efficacy of a Candida Vaccine in Women With Recurrent Vulvovaginal Candidiasis: A Randomized Controlled Study
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: LimmaTech Biologics AG (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Candi5V01; 2023-507527-28-00 (Other: CTIS)
Record Dates: First submitted 2023-12-19; First posted 2024-01-05 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Recurrent Vulvovaginal Candidiasis
Keywords: Recurrent Vulvovaginal Candidiasis; Vulvovaginal Candidiasis; Candida Vaccine
MeSH Terms: conditions — Candidiasis, Vulvovaginal | interventions — Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Candi5V half dose (Active Comparator)
  Interventions: Biological: Vaccine
- Candi5V half dose + adjuvant (Active Comparator)
  Interventions: Biological: Vaccine
- Candi5V target dose (Active Comparator)
  Interventions: Biological: Vaccine
- Candi5V target dose + adjuvant (Active Comparator)
  Interventions: Biological: Vaccine
- Placebo (Placebo Comparator)
  Interventions: Biological: Vaccine

INTERVENTIONS:
Biological: Vaccine — The candidate pentavalent bioconjugate vaccine (Candi5V) is administered twice, 2 months apart, with adjuvant.
  Arms: Candi5V half dose + adjuvant; Candi5V target dose + adjuvant
Biological: Vaccine — The candidate pentavalent bioconjugate vaccine (Candi5V) is administered twice, 2 months apart without adjuvant
  Arms: Candi5V half dose; Candi5V target dose
Biological: Vaccine — The placebo is administered twice, 2 months apart
  Arms: Placebo

SUMMARY:
In this study, the pentavalent bioconjugate candidate vaccine (Candi5V) against Candida will be tested to obtain first-time-in-human (FTIH) data on its safety, immunogenicity, and preliminary efficacy in women with recurrent vulvovaginal candidiasis.

DETAILED DESCRIPTION:
This is a First Time In Human (FTIH), phase I/II, double-blind, randomized, placebo-controlled study to evaluate the safety, immunogenicity and preliminary efficacy of the candidate pentavalent bioconjugate vaccine (Candi5V), administered twice, 2 months apart, with or without adjuvant.

The study will be conducted in two subsequent steps:

Step 1 (safety cohort): staggered enrolment of small groups of women with history of RVVC, sequentially administered with the half dose of Candi5V non-adjuvanted and with adjuvant or placebo, followed by groups administered with the target dose of Candi5V non-adjuvanted and with adjuvant or placebo.

Step 2 (target cohort): concurrent enrolment of women with history of RVVC, randomized 1:1:1 to Candi5V, Candi5V + adjuvant and placebo.

All study participants will be followed for 12 months after the second vaccination, to assess the vaccine safety profile, the immunological response and the recurrence of any VVC episode.

ELIGIBILITY:
Inclusion Criteria:

1. Good general health by medical history, laboratory findings and physical examination before receiving vaccination as judged by the Investigator.
2. Documented history of R-VVC, defined as 3 or more VVC episodes in the previous year, of which:

   1. at least 3 can be documented by a visit at a physician's office OR are documented by antifungal drug use as proven by a retrospective pharmacist drug delivery list, or electronic prescription by a physician
   2. at least one is culture OR microscopy confirmed (Pap smear, wet mount or Gram stain for Candida spp).

   Note: patients on chronic long-term treatment with documented RVVC diagnosis with at least 3 VVC episodes within the previous 3 years before enrolment, of which:
   1. at least 3 can be documented by a visit at a physician's office OR are documented by antifungal drug use as proven by a retrospective pharmacist drug delivery list, or electronic prescription by a physician
   2. at least one is culture OR lab-based microscopy confirmed for Candida spp (Pap smear, wet mount or Gram stain).

   may also be considered eligible if not on any antifungal treatment for at least 1-month preceding vaccination.
3. Participant who is willing and able to comply with the requirements of the protocol (e.g., completion of the study diary, return for follow-up visits).
4. Signed written informed consent obtained from the participant.
5. Females between 18-47 years (inclusive) of age at the time of the first vaccination practicing highly effective birth control from prior to first vaccination until at least 28 days after the last vaccination agreed by participants. Females between 48-50 years (inclusive) can be included if they are using combined (estrogen and progesteron containing) hormonal oral contraceptives from prior to first vaccination until at least 1 month after the last vaccination as agreed by participants.

Note: highly effective birth control is defined as a contraceptive method with failure rate of less than 1% per year when used consistently and correctly, in accordance with the product label. Examples of these include: combined (estrogen and progesteron containing) hormonal contraceptives associated with inhibition of ovulation (oral or intravaginal or transdermal); progesteron-only hormonal contraceptives associated with inhibition of ovulation (oral or injectable or implantable); intrauterine device; intrauterine hormone-releasing system (IUS); bilateral tubal occlusion; sexual abstinence; vasectomized partner (male partner sterilisation at least 6 months prior to the female participant's entry into the study, and if the relationship is monogamous.

Exclusion Criteria:

1. Health condition that, in the opinion of the Investigator, may interfere with optimal participation in the study or place the participant at increased risk of adverse events.
2. Acute disease including VVC-symptoms at the time of vaccination.
3. Any deviation from the normal range in biochemistry or haematology blood tests or urine safety laboratory clinically significant in the opinion of the Investigator.
4. Clinically significant abnormalities on physical examination.
5. Suspected or known hypersensitivity (including allergy) to any of the medicinal products or medical equipment whose use is foreseen in this study.
6. History of allergy to any vaccine.
7. Clinical conditions representing a contraindication to intramuscular vaccination and blood draws (e.g., coagulation disorder).
8. VVC therapy within 1 month preceding the 1st vaccination (participants meeting this criterion will be followed and may be re-screened at a later timepoint following a negative culture).
9. Participants with cervical diseases, or any other vulvovaginal conditions that may influence vaccine efficacy and VVC treatment.
10. Known or suspected impairment of immunological function, documented Human Immunodeficiency Virus (HIV) infection, asplenia/splenectomy, or history of autoimmune disease or lymphoproliferative disorder.
11. Positive blood test for HBsAg, HCV, HIV-1/2.
12. History of systemic administration of immunosuppressive drugs, i.e., corticosteroids, (PO/IV/IM) within the last month prior to 1st vaccination or for more than 14 consecutive days within 3 months prior to 1st vaccination, until the last blood sampling visit (i.e., prednisone or equivalent ≥20 mg/day). Inhaled and topical steroids are allowed.
13. Administration of antineoplastic and immune-modulating agents or chemotherapy within 3 months prior to informed consent.
14. Planned or actual administration of any licensed vaccine within 14 days prior to each vaccination and 30 days after each vaccination. Note: In case an emergency mass vaccination for an unforeseen public health threat is organized by the public health authorities, outside the routine immunization program, the time period described above can be reduced if necessary, for that vaccine provided it is licensed and used according to the local governmental recommendations and provided a written approval of the Sponsor is obtained.
15. Concurrently participating in another clinical study, at any time during the study period, in which the participant has been or will be exposed to an investigational or a non-investigational interventional vaccine/product (pharmaceutical product).
16. Body Mass Index (BMI) ≤19 and ≥30.
17. History of any chronic or progressive disease that according to judgment of the Investigator could interfere with the study outcomes or pose a threat to the participant's health.
18. Received an investigational or non-registered product (medicinal drug or vaccine), other than the study vaccine within 3 months prior to 1st administration of study vaccine, or planned use during the study period.
19. Administration of immunoglobulin and/or any blood products within the three months preceding the first dose of study vaccine.
20. Blood donation equal or greater to 500 mL of blood drawn within 3 months preceding the first vaccination or planned during the study period as reported by the participant.
21. Use of any systemic antibiotic therapy within 1 week preceding each vaccination.
22. Participants with an elective surgical intervention, planned during the study period until 28 days after 2nd vaccination.
23. Females lactating, pregnant, or intending to become pregnant as reported by the participant, within at least one month post second vaccination. Note: in case of unintended and unknown pregnancy from prior to first vaccination until at least 1 month after the last vaccination, pregnancy should be followed to term, any premature terminations should be reported, and the health status of the mother and child including date of delivery and the child's gender and weight should be reported after delivery.
24. Current and/or history of chronic alcohol consumption and/or drug abuse.
25. History of immune-mediated disease.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 251 (Estimated)
Dates: Start 2023-12-06 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
- Percentage of participants with solicited AEs at the administration site during the 7-day follow-up period (day of administration and 6 following days) after each dose, in the Candi5V arms and the placebo arm. | within 0-7 days after vaccination
- Percentage of participants with each solicited systemic AE during the 7-day follow-up period (day of administration and 6 following days) after each dose, in the Candi5V arms and the placebo arm. | within 0-7 days after vaccination
- Percentage of participants with unsolicited AEs during the 28-day follow-up period (day of administration and 27 following days) after each dose, in the Candi5V arms and the placebo arm. | within 0-28 days after vaccination
- Percentage of participants with SAEs from the first dose to study end in the Candi5V arms and the placebo arm. | up to 12 months after second vaccination
- Percentage of participants with medically relevant AEs from the first dose to study end. | up to 12 months after second vaccination
- Percentage of participants with AEs leading to withdrawal from the study or to the withholding of further study intervention administration, during their entire study participation, in the Candi5V arms and the placebo arm. | up to 12 months after second vaccination
- Percentage of participants with haematological and biochemical laboratory abnormalities at 7-days post-dose compared to pre-dose values (V3 vs V2, V7 vs V6) in the Candi5V arms and the placebo arm. | within 0-7 days after vaccination
- Percentage of participants with AESIs (e.g., pIMDs, vulvovaginal candidiasis, extravaginal candidiasis or systemic fungal infection) from the first dose to study end in the Candi5V arms and the placebo arm. | up to 12 months after second vaccination
- Evaluation of geometric mean titers (GMTs) for serum IgG against the five Candida antigens included in Candi5V, between baseline and post-vaccination samples collected at V8 (i.e., 28 days after the second vaccination). | within 0-28 days after vaccination

SECONDARY OUTCOMES:
- Evaluation of geometric mean titers (GMTs) for serum IgG against the five Candida antigens included in Candi5V, between baseline and post-vaccination samples collected at V5, in the Candi5V arms and the placebo arm. | within 0-28 days after vaccination
- Evaluation of geometric mean ratios (GMRs) for serum IgG against the five Candida antigens included in Candi5V, between baseline and post-vaccination (fold increase) on samples collected at V5 and V8, in the Candi5V arms and the placebo arm. | within 0-28 days after vaccination
- Percentage of participants in the Candi5V arms and the placebo arm achieving at least a four-fold rise (seroconversion) in the GMT of serum IgG against the Candi5V antigens at V5 and V8, compared to baseline. | within 0-28 days after vaccination
- Evaluation of geometric mean titers (GMTs) for serum IgA against the five Candida antigens included in Candi5V, between baseline and post-vaccination samples collected at V8, in the Candi5V arms and the placebo arm. | within 0-28 days after vaccination
- Evaluation of GMRs for serum IgA against the five Candida antigens included in Candi5V between baseline and post-vaccination (fold increase) on samples collected at V8, in the Candi5V arms and the placebo arm. | within 0-28 days after vaccination
- Percentage of participants in the Candi5V arms and the placebo arm achieving at least a four-fold rise (seroconversion) in the GMT of serum IgA against the Candi5V antigens at V8, compared to baseline. | within 0-28 days after vaccination
- Evaluation of GMTs for vaginal swab IgG and IgA against the five Candida antigens included in Candi5V between baseline and post-vaccination on samples collected at V8, in the Candi5V arms and the placebo arm. | within 0-28 days after vaccination
- Evaluation of GMRs for vaginal swab IgG and IgA against the five Candida antigens included in Candi5V between baseline and post-vaccination on samples collected at V8, in the Candi5V arms and the placebo arm. | within 0-28 days after vaccination
- Percentage of participants in the Candi5V arms and the placebo arm achieving at least a four-fold rise (seroconversion) in the GMT of vaginal swab IgG and IgA against the Candida antigens included in Candi5V at V8 compared to baseline. | within 0-28 days after vaccination
- Incidence rates of VVC cases during the 12 months post 2nd vaccination, in the Candi5V arms and the placebo arm. For the purpose of the case definition, only the first confirmed VVC infection will be considered. | up to 12 months after second vaccination
- Incidence rates of VVC cases from 28 days after 1st vaccination until end of the study, in the Candi5V arms and the placebo arm. For the purpose of the case definition, only the first confirmed VVC infection will be considered. | up to 12 months after second vaccination
- VVC recurrence rate during the 12 months post 2nd vaccination, in the Candi5V arms and the placebo arm. All infections experienced by the participants during the time of observation will be counted for this endpoint. | up to 12 months after second vaccination
- VVC recurrence rate from 28 days after the 1st vaccination until end of study, in the Candi5V arms and the placebo arm. All infections experienced by the participants during the time of observation will be counted for this endpoint. | up to 12 months after second vaccination
- Incidence rate of mild, moderate, or severe VVC during the 12 months post 2nd vaccination, in the Candi5V arms and the placebo arm. | up to 12 months after second vaccination
- Incidence rate of mild, moderate, or severe VVC 28 days after the 1st vaccination until end of study, in the Candi5V arms and the placebo arm. | up to 12 months after second vaccination
- As the above but for clinically confirmed VVC episodes independently on microscope and/or culture results. | up to 12 months after second vaccination
- Percentage of participants with extravaginal candidiasis or systemic fungal infection 28 days after the 1st vaccination to 12 months post 2nd vaccination, in the Candi5V arms and the placebo arm. | up to 12 months after second vaccination
- All efficacy endpoints will be analysed for any Candida spp and for C. albicans likewise. | up to 12 months after second vaccination

CONTACTS AND LOCATIONS:
Locations (6):
- Belgium (2):
  - Femicare, Tienen, Tienen
  - Universitair Ziekenhuis Gent, Ghent
- Poland (4):
  - Aidport sp.z o.o., Skórzewo, Poznan
  - IN-VIVO Sp. z o.o., Bydgoszcz
  - NZOZ Medem, Katowice
  - Velocity Nova sp. z o.o, Lublin

IPD SHARING:
Plan to Share IPD: No